CLINICAL TRIAL: NCT03491852
Title: Be Outspoken and Overcome Stigmatizing Thoughts: A Randomized Controlled Trial Targeting Self-Stigma in First Episode Psychosis
Brief Title: A Novel Treatment Approach for Self-Stigma in First Episode Psychosis
Acronym: BOOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Dr. Christopher Bowie, Principal Investigator, Professor, Deptartment of Psychology, Queen's University, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4077
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOOST Intervention (Experimental): The BOOST intervention consists of 8 group-based, weekly one-hour sessions. While every BOOST session is different, in general they will focus on helping participants fight back against stigmatizing thoughts and develop a sense of self-worth and empowerment. BOOST sessions are group-based and facilitated by trained clinicians, with the aid of a peer support worker to provide unique insights on living with and overcoming self-stigma. Content of sessions involve group discussions, exercises conducted in session, and between-session "missions" (i.e., home practice activities).
  Interventions: Behavioral: BOOST Intervention
- Waitlist Controls (Active Comparator): Participants on the waitlist will still receive treatment as usual, which includes medical, psychosocial, and occupational interventions to help maximize patients' integration within the community and support recovery from a first episode of psychosis. Frequency of contact largely depends on the individual needs of patients. Waitlist controls will be offered the BOOST intervention 3 months post-enrollment.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: BOOST Intervention — A cognitive and behavioural group therapy designed to reduce self-stigma and promote effective communication skills for adults (16-65 years old) experiencing a first episode of psychosis.
  Arms: BOOST Intervention
Behavioral: Waitlist Control — Participants on the waitlist will still receive treatment as usual, which includes medical, psychosocial, and occupational interventions to help maximize patients' integration within the community and support recovery from a first episode of psychosis.
  Arms: Waitlist Controls

SUMMARY:
Stigma towards mental illness is one of the greatest barriers to functional recovery that people with psychotic disorders face. Internalization of stigma (self-stigma) is associated with increased depressive symptoms, treatment non-adherence, and reduced quality of life. Self-stigma also has functional consequences, such as social avoidance and decreased help-seeking behaviour, which may worsen symptoms and impede recovery. Despite a growing awareness of the negative outcomes associated with self-stigma, few interventions have been designed to specifically address this experience in first episode psychosis. This project proposes to determine the effectiveness of an innovative, youth-oriented, group-based intervention known as Be Outspoken and Overcome Stigmatizing Thoughts (BOOST), which aims to reduce self-stigma and promote effective communication skills for adults (16-65 years old) experiencing a first episode of psychosis.

DETAILED DESCRIPTION:
BOOST is a manualized intervention that combines psychoeducation and cognitive restructuring to replace stigmatizing views about early psychosis and help patients challenge negative self-evaluations. Assertiveness skills training is a unique component that was added to the group to empower individuals and provide them with the behavioural skills to fight back against self-stigma and get their needs met during social interactions.

Sessions are 60 minutes long and occur once a week for 8 weeks. Groups comprise 4-6 outpatients enrolled in a specialized outpatient clinic for early psychosis. Session are led by one therapist and co-facilitated with a peer support worker who has "lived experience" with early psychosis to provide unique insights on living with and overcoming self-stigma. The group format is informal and discussion-based, with an emphasis on sharing personal experiences.

Early sessions (1-4) focus on dispelling popular myths associated with psychosis and challenging erroneous beliefs, as a way to provide psychoeducation to patients. Additionally, time is spent identifying the impact of self-labelling, how this can lead to self-fulfilling prophecies, and getting participants to reflect on examples of when self-stigma might have behavioural consequences. Cognitive behavioural therapy techniques are used as a basis for the intervention, with an initial focus on cognitive restructuring to fight back against negative, stigmatizing thoughts.

Later sessions (5-8) target behavioural approaches for self-empowerment through assertiveness skills training and goal setting. Discussions are focused on the verbal and non-verbal characteristics of passive, aggressive, and assertive communication, in addition to techniques for speaking in an assertive manner. Role play scenarios that are specific to young people with psychosis provide opportunities to practice these skills in session. For example, Speaking up to a psychiatrist about the negative side effects of a medication or reaching out to a friend for support after returning from a hospitalization.

Weekly "missions" (i.e., home practice activities) are administered following each session to build on group content and help participants fight back against self-stigmatizing thoughts and attitudes in everyday contexts.

ELIGIBILITY:
Inclusion Criteria:

* Involvement in an early psychosis clinic for a period of less than 3 years, due to the focus of this study being on the treatment of early psychosis. Participants must be between the ages of 16 and 65 years. Participants 16 years of age who are incapable to consent without a parent or guardian will be excluded. Participants must be fluent in English, as determined by referring clinicians or researchers (in the case of advertisement referred participants) in order to meaningfully participate in the BOOST intervention and complete the assessment tools.

Exclusion Criteria:

* Potential participants who are unable to provide informed consent, as determined by the treatment team, will not be able to meaningfully participate in the BOOST intervention and will, therefore, be unable to participate in the research study. Individuals with a presence of intellectual disability or history of traumatic brain injury will also be excluded.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Stigma - Internalized Stigma of Mental Illness Scale (ISMI) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  The ISMI (Ritsher, Otilingam, & Grajales, 2003) is a 29-item self-report questionnaire designed to assess subjective experience of stigma.

SECONDARY OUTCOMES:
Change in Self-Esteem - Rosenberg Self-Esteem Scale (RSES) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  The RSES (Rosenberg et al., 1995) is a 10-item self-report questionnaire that IS used to measure self-esteem.
Change in Quality of Life - Satisfaction with Life Safe (SWLS) from Baseline | Post-treatment (within 2 weeks following the end of treatment)
  The SWLS (Kobau et al., 2010) is a short 5-item instrument designed to measure global cognitive judgments of satisfactions with one's life.
Change in Stigma Stress - Cognitive Appraisal of Stigma Stress (CogApp) | Post-treatment (within 2 weeks following the end of treatment)
  The CogApp (Rüsch et al., 2009) is an 8-item measure that yields a difference score of stigma stress by subtracting perceived resources to cope with stigma from perceived stigma-related harm.
Change in Depression - Beck Depression Inventory-II (BDI) | Post-treatment (within 2 weeks following the end of treatment)
  The BDI-II (Beck, Steer, & Brown, 1996) is a 21-item self-report instrument intended to assess the existence and severity of symptoms of depression.
Change in Social Anxiety - Social Interaction Anxiety Scale (SIAS) | Post-treatment (within 2 weeks following the end of treatment)
  The SIAS (Mattick & Clarke, 1998) is a 20 item self-report scale designed to measure social interaction anxiety.
Change in Personal Recovery - Questionnaire about the Process of Recovery (QPR) | Post-treatment (within 2 weeks following the end of treatment)
  The QPR (Williams et al., 2015) is a 22-item, service user-rated measure of personal recovery.
Change in Functioning - Sheehan Disability Scale (SDS) | Post-treatment (within 2 weeks following the end of treatment)
  The SDS (Sheehan et al., 1996) is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowie, PhD, Principal Investigator — Queen's University
Locations (1):
- St. Joseph's Healthcare Hamilton, West 5th Campus, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No